CLINICAL TRIAL: NCT04295785
Title: Clinical, Paraclinical, Functional Characteristics and Evolution of Juvenile Autoimmune Necrotizing Myopathies in a National Retrospective Cohort
Brief Title: Juvenile Autoimmune Necrotizing Myopathies
Acronym: MYONECPED
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI192
Record Dates: First submitted 2020-01-09; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-01

CONDITIONS: Immune-Mediated Necrotizing Myopathy
Keywords: Autoimmune necrotizing myopathy; anti-HMGCR antibodies; anti-SRP antibodies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- autoimmune necrotizing myopathy beginning before 18

SUMMARY:
Autoimmune necrotizing myopathies (AINM) in adult patients are characterized by severity of muscle damage, presence of necrosis with little inflammation on muscle biopsy and anti-HMGCR or anti-SRP auto-antibodies. Data on AINM in children are currently lacking. The purpose of this study is to specify the characteristics at AINM diagnosis, treatments and evolution of juvenile AINM with anti-HMGCR or anti-SRP antibodies.

ELIGIBILITY:
Inclusion Criteria:

* AINM histologically proved by predominant muscle fibers necrosis lesions associated with minimal or absent inflammatory lesions
* Either anti-SRP or anti-HMGCR antibodies positivity
* Disease onset before age 18

Exclusion Criteria:

* Seronegative necrotizing myopathies
* Forms compatible with another type of myositis (e.g. dermatomyositis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: AINM histologically proved (i.e. predominant muscle fibers necrosis lesions associated with minimal or absent inflammatory lesions), either anti-SRP or anti-HMGCR antibodies positivity and a disease onset before age 18
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Type of muscle involvment | At diagnosis
  Proximal or distal or axial muscle involvement by muscle testing
Type of cutaneous involvment | At diagnosis
  Rash or Gottron lesions
Other clinical manifestations | At diagnosis
  Dysphagia or dyspnea or fever or interstitial lung involvement or articular involvement or gastrointestinal involvment
Blood CK level | At diagnosis
  Blood CK level
Histology | At diagnosis
  Results of muscle biopsy : necrosis
Histology | At diagnosis
  Results of muscle biopsy : inflammation
MMT score | At diagnosis
  MMT score
CMAS score | At diagnosis
  CMAS score

SECONDARY OUTCOMES:
Type of drugs used | At last visit
  Drugs ever used : name and duration
Iatrogenic complications | At last visit
  Infectious complications
Iatrogenic complications | At last visit
  Bone complications
Status of the disease at last visit | At last visit
  Status of the disease at last visit : active or remission or death
Number of relapses | At last visit
  Number of relapses
Type of muscle involvment | At last visit
  Proximal or distal or axial muscle involvement by muscle testing
Type of cutaneous involvment | At last visit
  Rash or Gottron lesions
Other clinical manifestations | At last visit
  Dysphagia or dyspnea or fever or interstitial lung involvement or articular involvement or gastrointestinal involvment
Blood CK level | At last visit
  Blood CK level
CMAS score | At last visit
  CMAS score
MMT score | At last visit
  MMT score

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital d'enfants CHRU Nancy, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Background] Benveniste O, Stenzel W, Allenbach Y. Advances in serological diagnostics of inflammatory myopathies. Curr Opin Neurol. 2016 Oct;29(5):662-73. doi: 10.1097/WCO.0000000000000376. PMID 27538058
- [Background] Mariampillai K, Granger B, Amelin D, Guiguet M, Hachulla E, Maurier F, Meyer A, Tohme A, Charuel JL, Musset L, Allenbach Y, Benveniste O. Development of a New Classification System for Idiopathic Inflammatory Myopathies Based on Clinical Manifestations and Myositis-Specific Autoantibodies. JAMA Neurol. 2018 Dec 1;75(12):1528-1537. doi: 10.1001/jamaneurol.2018.2598. PMID 30208379
- [Background] Watanabe Y, Uruha A, Suzuki S, Nakahara J, Hamanaka K, Takayama K, Suzuki N, Nishino I. Clinical features and prognosis in anti-SRP and anti-HMGCR necrotising myopathy. J Neurol Neurosurg Psychiatry. 2016 Oct;87(10):1038-44. doi: 10.1136/jnnp-2016-313166. Epub 2016 May 4. PMID 27147697
- [Background] Allenbach Y, Drouot L, Rigolet A, Charuel JL, Jouen F, Romero NB, Maisonobe T, Dubourg O, Behin A, Laforet P, Stojkovic T, Eymard B, Costedoat-Chalumeau N, Campana-Salort E, Tournadre A, Musset L, Bader-Meunier B, Kone-Paut I, Sibilia J, Servais L, Fain O, Larroche C, Diot E, Terrier B, De Paz R, Dossier A, Menard D, Morati C, Roux M, Ferrer X, Martinet J, Besnard S, Bellance R, Cacoub P, Arnaud L, Grosbois B, Herson S, Boyer O, Benveniste O; French Myositis Network. Anti-HMGCR autoantibodies in European patients with autoimmune necrotizing myopathies: inconstant exposure to statin. Medicine (Baltimore). 2014 May;93(3):150-157. doi: 10.1097/MD.0000000000000028. PMID 24797170
- [Background] Anti-HMGCR Autoantibodies in Juvenile Idiopathic Inflammatory Myopathies Identify a Rare but Clinically Important Subset of Patients. J Rheumatol. 2017 Sep;44(9):1417. doi: 10.3899/jrheum.160871.C1. No abstract available. PMID 28864670
- [Background] Liang WC, Uruha A, Suzuki S, Murakami N, Takeshita E, Chen WZ, Jong YJ, Endo Y, Komaki H, Fujii T, Kawano Y, Mori-Yoshimura M, Oya Y, Xi J, Zhu W, Zhao C, Watanabe Y, Ikemoto K, Nishikawa A, Hamanaka K, Mitsuhashi S, Suzuki N, Nishino I. Pediatric necrotizing myopathy associated with anti-3-hydroxy-3-methylglutaryl-coenzyme A reductase antibodies. Rheumatology (Oxford). 2017 Feb;56(2):287-293. doi: 10.1093/rheumatology/kew386. Epub 2016 Nov 6. PMID 27818386
- [Background] Tiniakou E, Pinal-Fernandez I, Lloyd TE, Albayda J, Paik J, Werner JL, Parks CA, Casciola-Rosen L, Christopher-Stine L, Mammen AL. More severe disease and slower recovery in younger patients with anti-3-hydroxy-3-methylglutaryl-coenzyme A reductase-associated autoimmune myopathy. Rheumatology (Oxford). 2017 May 1;56(5):787-794. doi: 10.1093/rheumatology/kew470. PMID 28096458
- [Background] Binns EL, Moraitis E, Maillard S, Tansley S, McHugh N, Jacques TS, Wedderburn LR, Pilkington C, Yasin SA, Nistala K; UK Juvenile Dermatomyositis Research Group (UK and Ireland). Effective induction therapy for anti-SRP associated myositis in childhood: A small case series and review of the literature. Pediatr Rheumatol Online J. 2017 Oct 31;15(1):77. doi: 10.1186/s12969-017-0205-x. PMID 29089059